CLINICAL TRIAL: NCT06785233
Title: Endoscopic Treatment of Overweight and Mild Obesity Using a 12-month Non-adjustable Intragastric Balloon (ORBERA365)
Brief Title: Endoscopic Treatment of Overweight and Mild Obesity with ORBERA365
Acronym: ORBERA365
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Clinic and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISR ORBERA365
Record Dates: First submitted 2025-01-09; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Obesity, Morbid
Keywords: obesity; Intragastric Balloon
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: endoscopic treatment of overweight and mild obesity using a 12-month non-adjustable intragastric balloon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intragastric Ballon (Experimental): Endoscopic placement of Orbera365® non-adjustable intragastric balloon under general anesthesia. Device filled with 600mL saline solution with methylene blue, remaining in situ for 12 months. Weekly follow-up in first month, then monthly visits including nutritional and psychological support. Removal performed under general anesthesia after 12-month period.
  Interventions: Device: Non-Adjustable Intragastric Balloon; Device: ORBERA365

INTERVENTIONS:
Device: Non-Adjustable Intragastric Balloon — Weight Loss with a 12-Month Non-Adjustable Intragastric Balloon is More Effective Compared to a 6-Month Balloon.
Device: ORBERA365 — endoscopic treatment of overweight and mild obesity using a 12-month non-adjustable intragastric balloon
  Other Names: Intragastric Balloon

SUMMARY:
INTRODUCTION: Obesity is a critical health condition associated with high rates of morbidity and mortality. Conservative therapies such as dietary restriction, physical exercise, and pharmacological treatments have not prevented the rising incidence of obesity. Bariatric surgery, while effective, is limited to a relatively small proportion of the global obese population due to its strict indications and the risk of early and late postoperative complications. To address this gap, bariatric endoscopy therapies have emerged, offering less invasive, reversible, repeatable, and more cost-effective treatment options. The introduction of the intragastric balloon (IGB) in the 1980s marked the development of a minimally invasive, non-surgical, and safe procedure with low complication rates. OBJECTIVE: To evaluate the weight loss efficacy in overweight and Class I obese patients through the implantation of a 12-month non-adjustable intragastric balloon. METHODS: This prospective study involved overweight patients (BMI > 27 kg/m²) undergoing intragastric balloon treatment and multidisciplinary follow-up at the Bariatric Endoscopy Clinic of the Faculty of Medicine of ABC (FMABC) over a 12-month period. EXPECTED RESULTS: Weight loss following intragastric balloon implantation and improvement in metabolic indices.

DETAILED DESCRIPTION:
Research Objective: The primary objective of this research will be to evaluate weight loss in overweight or class I obesity patients following the implantation of the Orbera365® non-adjustable intragastric balloon. The secondary objective will be to correlate demographic, endoscopic, and laboratory data with the outcomes of this procedure.

Patients and Methods: Patients with BMI > 27 kg/m² or BMI between 30-35 kg/m², regardless of gender and ethnic background, will undergo Orbera365® intragastric balloon implantation. The procedures will be performed at the Endoscopy Service of Mario Covas Hospital in São Paulo, SP and Kaiser Clinic in São José do Rio Preto, SP. Data collection will be conducted at the same locations. Information will be obtained during outpatient follow-up, including demographic data (sex, age), clinical data (height, weight, metabolic comorbidities), and operative data (complications).

Procedure Preparation: All examinations will be performed following a minimum 8-hour fasting period. The procedure will be initiated with the patient in left lateral decubitus under general anesthesia administered by an anesthesiologist. The balloon will be implanted under direct visualization in the gastric fundus and filled with up to 600 mL of 0.9% saline solution and 2% methylene blue.

Post-Procedure Recovery: Following the procedure and anesthesia recovery, all patients will be discharged but only with an accompanying person. All patients will receive guidance and will maintain contact with a physician to report any adverse signs or symptoms. Follow-up will include weekly consultations during the first month and monthly consultations thereafter, totaling one year of monitoring.

Outcomes: Primary outcome: To confirm the efficacy of the Orbera365® intragastric balloon in the primary treatment of obesity through evaluation of total weight loss.

Secondary outcome: To evaluate the use of the intragastric balloon in relation to demographic data and its impact on metabolic comorbidities.

Statistical Analysis: Analysis will be performed using Minitab Statistical Software, including normality tests, comparisons between numerical variables (Student's t-test or Mann-Whitney) and categorical variables (Pearson's chi-square or Fisher's exact test), considering p < 0.05 as significant.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a Body Mass Index (BMI) above 27 kg/m²,
* both sexes,
* aged 18 years or older,
* who consent to their participation by signing an Informed Consent Form and
* agree to the implantation of the Orbera365® balloon at Kaiser Clinic and the Faculty of Medicine of ABC (FMABC)/Hospital Mario Covas.

Exclusion Criteria:

* Relative or absolute contraindications for this procedure, such as hiatal hernia (> 3 cm),
* Los Angeles grade erosive esophagitis,
* peptic ulcer,
* prior gastric surgery,
* substance dependence (alcohol or illicit drugs),
* continuous anticoagulant or anti-inflammatory therapy, and those with
* positive urease test results until treatment is completed and evidence of resolution is provided or follow-up is lost.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Orbera365® intragastric balloon. | 12 weeks
  Weight loss following the implantation of the Orbera365® intragastric balloon.
  Weight loss following the implantation of the Orbera365® intragastric balloon. Weight loss following the implantation of the Orbera365® intragastric balloon.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Luiiz Kaiser Junior, Study Chair — Kaiser Clinica
Locations (1):
- Faculdade ABC, Santo André, São Paulo, Brazil